CLINICAL TRIAL: NCT03281460
Title: Efficacy of In-bag Morcellation
Acronym: FIBROSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0714; 2017-A01773-50 (Other: ID-RCB)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Uterine Myomatosis; Laparoscopy; Hysterectomy, Vaginal
Keywords: Hysterectomy, Vaginal; Uterine Myomatosis; Morcellation; Laparoscopy; in-bag morcellation
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with in-bag morcellation (Experimental): with More-cell-Safe AMI bag morcellation
  Interventions: Device: laparoscopic myomectomy or hysterectomy with More-cell-Safe AMI bag morcellation
- without any morcellation bag (Active Comparator): without any morcellation bag
  Interventions: Procedure: laparoscopic myomectomy or hysterectomy without any morcellation bag

INTERVENTIONS:
Device: laparoscopic myomectomy or hysterectomy with More-cell-Safe AMI bag morcellation — laparoscopic myomectomy or hysterectomy with More-cell-Safe AMI bag morcellation
  Arms: with in-bag morcellation
Procedure: laparoscopic myomectomy or hysterectomy without any morcellation bag — laparoscopic myomectomy or hysterectomy without any morcellation bag
  Arms: without any morcellation bag

SUMMARY:
Laparoscopic mini-invasive surgery supplanted laparotomy for many years, including hysterectomy or myomectomy (less postoperative complications compared to laparotomy) However the US Federal Drug Administration (FDA) strongly warned against the use of power morcellation in 2014 because of the risk of iatrogenic spread of malignant cells.

The hypothesis is that in-bag morcellation may prevent cells dissemination. The investigator compare in this prospective randomized study two groups of patients: group A (in bag-morcellation during laparoscopic myomectomy or hysterectomy) versus group B (morcellation without any bag during laparoscopic myomectomy or hysterectomy)

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or more
* Laparoscopic myomectomy or laparoscopic subtotal hysterectomy
* Informed and signed consent

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* Preoperative risk of leiomyosarcoma or pelvic carcinoma
* Pregnancy or desire of pregnancy during the study period
* Uterus or myomas weight above 1.000 g
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Smooth muscular cells in the peritoneal fluid after morcellation | Day 0 - just after surgery
  After morcellation, there will be cytology and immunohistochemistry of peritoneal washing with 500cc of saline serum

SECONDARY OUTCOMES:
duration of surgery | Day 0
morcellation time | Day 0 - during surgery
peritoneal washing time | Day 0 - during surgery
residual morcellated tissues weight | Day 0 - during surgery
bag associated time | Day 0 - during surgery
ease of use | Day 0 - during surgery
  assessment by a visual analogical scale

CONTACTS AND LOCATIONS:
Overall Officials: Gautier CHENE, MD, Principal Investigator — Gynaecology Department, Hôpital Femme Mère Enfant, HCL
Locations (1):
- Gynaecology Department, Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bensouda-Miguet C, Nohuz E, Cerruto E, Buenerd A, Nadaud B, Moret S, Chene G. Inbag Morcellation Applied to the Laparoscopic Surgery of Leiomyoma: A Randomized Controlled Trial. Biomed Res Int. 2021 May 26;2021:6611448. doi: 10.1155/2021/6611448. eCollection 2021. PMID 34136570